CLINICAL TRIAL: NCT05761587
Title: Validation of a Screening Scale for the Misuse of Opioid Analgesics in Patients With Chronic Pain Related to Cancer.
Brief Title: Validation of a Screening Scale for Misuse of Opioid Analgesics
Acronym: VPOMIONCOL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2022 GUASTELLA
Record Dates: First submitted 2023-02-16; First posted 2023-03-09 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-02

CONDITIONS: Cancer; Pain; Opioid Analgesic Adverse Reaction
MeSH Terms: conditions — Neoplasms; Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cancer patients: Questionnaires
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — questionnaire including socio-demographic data, medical and family history, lifestyle, treatments, 5 questions from the Questionnaire Concis sur les Douleurs (QCD), the French version of the POMI scale, the diagnostic criteria of the DSM-V and two questions concerning anxiety associated with pain and therapeutic education.

SUMMARY:
In oncology, pain is one of the main symptoms of discomfort. It has a significant impact on the quality of life.The use of opioid analgesics is recommended for the treatment of moderate to severe cancer pain.The misuse of opioid analgesics is an international public health problem.Different scales have been developed to help the prescriber screen for the risk of misuse in the general population. Patients with cancer-related pain are also at risk for aberrant opioid-related behaviors, misuse or addiction.

The main objectif of this study is to validate of the screening scale for the misuse of opioid analgesics in patients with chronic pain related to cancer. (Prescription Opioid Misuse Index - POMI).

DETAILED DESCRIPTION:
The study takes place in 2 phases.

Test phase :

Questionnaire no. 1 constitutes the data for the TEST phase: it includes socio-demographic data, medical and family history, lifestyle, treatments, 5 questions from the Concise Pain Questionnaire (QCD), the French version of the POMI scale, the diagnostic criteria of the DSM-V and two questions concerning anxiety associated with pain and therapeutic education.

Retest phase :

questionnaire no. 2 10 to 15 days later.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over,
* Patients with chronic cancer-related pain that has been evolving for at least 3 months,
* Patients with a regular prescription of at least one opioid analgesic medicine taken daily for at least 1 month,
* Patients followed in oncology for an active cancerous pathology.

Exclusion Criteria:

* Stopping opioid prescriptions on the day of the test phase (no Retest possible),
* Patients in the process of weaning (risk of being weaned during the Retest phase),
* Patients unable to complete the questionnaire on their own,
* Patients followed in a pain or addiction centre,
* Patients in terminal palliative situations of their cancer,
* Patients with chronic pain that is more disabling than cancer-related pain,
* Patients refusing to participate,
* Patients under guardianship or curatorship,
* Pregnant or breastfeeding patients,
* Patient with a language barrier limiting understanding of the questionnaire in French.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
POMI scale score - Prescription Opioid Misuse Index | day 1
  8-item self-assessment scale
POMI scale score - Prescription Opioid Misuse Index | day 15
  8-item self-assessment scale

SECONDARY OUTCOMES:
QCD | day 1
  Visual Analogue Scales (VAS) for assessing the intensity and daily impact of pain (0-10)
QCD | day 15
  Visual Analogue Scales (VAS) for assessing the intensity and daily impact of pain (0-10)
Sociodemographic characteristics | day 1
  Questionnaire about Sociodemographic characteristics of patients
Lifestyle habits, other consumption | day 1
  Questionnaire about Lifestyle habits, other consumption
Analgesic treatments | day 1
  Questionnaire about Ongoing analgesic treatments
Use of analgesics | day 1
  Question evaluating the use of analgesics in the context of anticipating pain
Use of analgesics | day 15
  Question evaluating the use of analgesics in the context of anticipating pain

CONTACTS AND LOCATIONS:
Overall Officials: Virginie Guastella, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (2):
- France (2):
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CH Le Puy en Velay, Le Puy-en-Velay